CLINICAL TRIAL: NCT02379286
Title: Impact of Media Images, Alcohol and Tobacco to youthImpact Study and Development of a Prevention Program
Brief Title: Impact of Media Images, Alcohol and Tobacco to Youth
Acronym: IMAJE
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-02
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
MeSH Terms: interventions — Contact Tracing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 14 to 17 years old French teenager: 14 to 17 years old French teenager representative of French population from whom parental consent to particpare to the study has been given
  Interventions: Other: Investigation

INTERVENTIONS:
Other: Investigation — Investigation of relationships between French teenagers' attitudes and beliefs towards alcohol and tobacco products and the degree to which they watch and relate to television series and music videos

SUMMARY:
The main objective is to assess the relationships between French teenagers' attitudes and beliefs towards alcohol and tobacco products and the degree to which they watch and relate to television series and music videos.

DETAILED DESCRIPTION:
The research extends existing research conducted by Cristel A. Russell to assess the relationships between French teenagers' attitudes and beliefs towards alcohol and tobacco products and the degree to which they watch and relate to television series and music videos. We test whether the consumption of media (TV series and music video) are related to French youth's perceptions of the consequences related to the use of alcohol and/or tobacco and ultimately their intentions and behaviors. To do so, an online questionnaire will be passed. Teenagers will be recruited through a private research firm, Cint. Because the study focuses on teenagers (14-17 y.o), parental consent to participate to the study will be obtained prior to the teenager's one.

ELIGIBILITY:
Inclusion Criteria:

* Ages between14 to 17 years inclusive;
* Have access to television

Exclusion Criteria:

* Refusal to participate

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Tennagers aged between 14 and 17 years
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Connectedness scale to media and intention of drinking and/or smoking | 15 minutes
  Connectedness scale to media and intention of drinking and/or smoking

CONTACTS AND LOCATIONS:
Overall Officials: Franck Chauvin, PhDMD, Study Director — ICLN